CLINICAL TRIAL: NCT05587010
Title: Comparison of Gait in Different Support Conditions for Foot Drop
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr Tim Exell (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government); Solent NHS Trust (Other Government)
Responsible Party: Sponsor-Investigator, Dr Tim Exell, Senior Lecturer inn Biomechanics and Rehabilitation Science, University of Portsmouth
Organization: University of Portsmouth (Other)
Other Study IDs: Orthoped-UoP-22
Record Dates: First submitted 2022-10-11; First posted 2022-10-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Foot Drop, Unspecified Foot
Keywords: orthotic; AFO
MeSH Terms: conditions — Peroneal Neuropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Foot drop: Participants living with foot drop in either foot. Orthotic support devices will be compared within this cohort to assess their impact on gait biomechanics and clinical outcomes
  Interventions: Device: AFO; Device: lycra sock; Device: OrthPed splint

INTERVENTIONS:
Device: AFO — ankle foot orthosis
Device: lycra sock — custom fitted lycra sock
Device: OrthPed splint — novel compression splint

SUMMARY:
Foot drop is a complication accompanying a variety of conditions and refers to difficulty in lifting the foot upwards about the ankle. Foot drop is a common outcome of conditions including cerebral palsy, brain/spinal cord injury, muscular dystrophy, stroke and after chemotherapy. Foot drop can lead to trips and falls for the individual if the foot catches on the ground when walking, negatively impacting on independence and quality of life.

Approximately 46,720 children and adolescents in the UK have the above conditions and current treatment for individuals with foot drop include use of a lycra sock for those requiring low support and a rigid Ankle Foot Orthosis (AFO) for those requiring high support. The current problem is that all children and adolescents requiring more than low support of the lycra sock are fitted with an AFO, which can lead to muscles becoming weak over time as the AFO restricts almost all movement about the ankle.

This study will assess the use of a new device, the OrthoPed splint, in young people aged 4 - 17 years old who have moderate foot drop. The OrthoPed splint has been developed to be used as a long-term device and aims to reduce loss of strength by allowing more ankle function than an AFO.

This study aims to assess the feasibility of recruiting children and adolescents with foot drop into a study, collecting information on their movement and how well they walk when wearing different support devices for foot drop. Each person in the study will be measured when walking barefoot (no external support) and when wearing an AFO, Lycra sock and the OrthoPed splint. This feasibility study will inform the design, management, and delivery of a future larger randomised, controlled, non-inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 - 17 years old
* Diagnosed moderate unilateral or bilateral foot drop
* Able to walk independently
* Minimum of 5 degrees of ankle dorsiflexion with or without gravity (Oxford Scale 2-4, Clarkson (2010))

Exclusion Criteria:

* Younger than 4 or older than 17 years old
* Severe foot drop that requires higher levels of support than elastic splint
* Unable to walk independently
* Visual impairment when corrected to not be able to see targets when walking
* Unable to understand and or cooperate with study protocol
* Health contraindications to exercise e.g. cardiac disease

Ages: 4 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Patients under paediatric physiotherapy care suffering from moderate foot drop. Patients will be identified through physiotherapy care for foot drop. As the OrthoPed splint is designed for use with moderate foot drop patients, we will only study patients identified by the physiotherapy team as having moderate foot drop, defined as a minimum of 5 degrees of dorsiflexion with or without gravity (Oxford Scale 2-4), and suitable for using the OrthoPed splint. The splint is aimed for use in children and adolescents aged between 2 - 17 Years but due to the need to follow instructions and understand the requirements of the study, we will only study children and adolescents aged 4-17 Years.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment as defined by the proportion of people with foot drop accepting the invitation to take part in the study | 6 months

SECONDARY OUTCOMES:
Joint angles during walking gait | 6 months
  Differences in peak flexion, extension and range of motion of ankle, knee, hip and elbow angles during walking gait in different support conditions
Step length during walking gait | 6 months
  Differences in step length in different support conditions
Step frequency during walking gait | 6 months
  Differences in step frequency in different support conditions
Step velocity during walking gait | 6 months
  Differences in step velocity in different support conditions
Ground reaction force during walking gait | 6 months
  Differences in peak vertical, anterior, posterior, medial and lateral ground reaction forces during walking gait in different support conditions
Parent reported outcome measures of gait comfort and capacity | 6 months
  Family Impact Module of Pediatric Quality of Life Inventory (PedsQL) (Varni et al. (2005)
Patient reported outcome measures of gait comfort and capacity | 6 months
  Core Module of PedsQL (Varni et al. (2005) in different support conditions
Distance walked during 6-minute walk test | 6 months
  Distance walked during 6-minute walk test in different support conditions
Time achieved during Single Leg Stand test | 6 months
  Time achieved during Single Leg Stand test in different support conditions
Time achieved during Timed Up and Go test | 6 months
  Time achieved during Timed Up and Go test in different support conditions
Score achieved from Gait Assessment and Intervention Tool | 6 months
  Score achieved from Gait Assessment and Intervention Tool in different support conditions
Time taken to put on each device 1 handed | 6 months
  Time taken to put on each device 1 handed

CONTACTS AND LOCATIONS:
Locations (1):
- University of Portsmouth, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
processed outcome results will be shared through dissemination and publication of results